CLINICAL TRIAL: NCT07396896
Title: Single-arm, Open-label, Single-center, Non-profit Interventional Clinical Trial on the Effects of the Ketogenic Diet in Patients With Brain Tumors and Central Obesity
Brief Title: KETO-TUMOR: a Study on Brain Tumors and Central Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Iacopo Sardi, MD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KETO-TUMOR
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obese Patients; Hypothalamic Neoplasms
MeSH Terms: conditions — Hypothalamic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keto-tumor (Experimental)
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Atkins Modified Diet (MAD)

SUMMARY:
Hypothalamic-chiasmatic tumours account for 5-10% of CNS tumours in children and can compromise hypothalamic function, causing alterations in energy balance and weight gain. In inoperable cases, chemotherapy and radiotherapy are used; the latter, although the gold standard, is associated with significant neurocognitive and endocrine-metabolic side effects, proportional to the hypothalamic damage.

The ketogenic diet, used for decades in the treatment of drug-resistant childhood epilepsy, induces the use of ketone bodies as a source of energy for the brain and is effective in controlling seizures. Among the different variants, the modified Atkins diet was chosen in this study to promote better patient adherence.

This study aims to evaluate the effectiveness of the ketogenic diet (KD) in treating central obesity secondary to hypothalamic-chiasmatic tumours (gliomas, craniopharyngiomas, germ cell tumours, etc.), which often lead to excessive weight gain. This is refractory to drug therapy and lifestyle changes, such as low-calorie diets and exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hypothalamic-chiasmatic tumour according to the WHO 2021 classification
2. Diagnosis of hypothalamic obesity: after 5 years of age, BMI >97th percentile in the WHO 2007 curves
3. Males and females aged between 7 and 30 years
4. Performance status: Lansky score > 40 for patients aged < 18 years and Karnofsky score > 40 for patients aged between 18 and 30 years
5. Signature of informed consent to participate in the study
6. Signature of consent by the minor patient to participate in the study (7-13 years and 14-17 years).

Exclusion Criteria:

1. Deficiencies of:

* Primary carnitine
* Carnitine palmitoyltransferase 2 (CPT 2)
* Carnitine acylcarnitine translocase (CACT)
* Beta-oxidation
* Medium-chain acyl-CoA dehydrogenase (MCAD)
* long-chain acyl-CoA dehydrogenase (LCAD)
* short-chain acyl-CoA dehydrogenase (SCAD)
* porphyria
* pyruvate carboxylase
* long-chain 3-hydroxyacyl-CoA dehydrogenase.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who experience weight loss of at least 5% over 24 months | From enrollment to the end of the follow up period at 24 months

SECONDARY OUTCOMES:
Percentage of patients showing weight reduction, improvement in lipid and carbohydrate parameters | From enrollment to the end of the follow up period at 24 months
Percentage of patients with ketosis | From enrollement to the end of the follow up period at 24 months
Percentage of patients with serious adverse events | From enrollement to the end of the follow up period at 24 months
Adherence rate to the proposed dietary intervention, considering the number of patients who discontinue the diet and those who continue it | From enrollment to the end of the follow up at 24 months
Percentage of patients showing reduction of lean body mass in 24 months | From enrollment to the end of the follow up period at 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No